CLINICAL TRIAL: NCT02711774
Title: Changes in Optic Nerve Sheath Diameter in Response to Various Levels of End Tidal Carbon Dioxide Levels in Healthy Patients Under General Anaesthesia
Brief Title: Changes in Optic Nerve Sheath Diameter in Response to Various Levels of End Tidal Carbon Dioxide Levels
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Indu Kapoor, Assistant Professor, All India Institute of Medical Sciences
Other Study IDs: IEC-128/05.02,2016, RP-34/2016
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Brachial Plexus Injury
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ultrasonography — ONSD will be measured by a 6-13 MHz linear probe of the ultrasound machine.

SUMMARY:
Intracranial Pressure ( ICP ) monitoring is an essential component of traumatic brain injured ( TBI ) patients management. The clinical signs of raised ICP may be unreliable and may reflect relatively late cerebral decompensation. ICP may be monitored by invasive or non invasive techniques. While invasive techniques show the real time values of ICP, they are associated with many complications like, intracranial bleeding and infection, occlusion of the catheter tip by blood, debris and difficult to locate ventricle in presence of cerebral oedema. All these drawbacks of invasive methods can be averted by employing non invasive techniques of ICP monitoring. Although they do not show a real time value but are excellent tools to detect presence or absence of raised ICP. Elevated ICP can be detected by Computarised tomographic scan (CT) or Magnetic resonance imaging (MRI) but , these techniques are time consuming and require transportation of a patients who may be unstable .The quick and non invasive nature of ultrasonography is fast becoming popular for rapid detection of elevated ICP at bedside in emergency and ICU by monitoring the optic nerve sheath diameter ( ONSD ). Its limitations notwithstanding, ultrasonographic ONSD monitoring is likely to be more reliable than clinical assessment in the diagnosis of intracranial hypertension especially, when patient is under sedation which precludes proper clinical examination. Therefore, in recent years ,among non invasive methods, bedside ocular ultrasonography to monitor ICP has gained popularity.

Carbon dioxide being a potent modulator of cerebral vascular tone, alters the ICP by changing the size of cerebral vasculature and thereby, cerebral blood flow (CBF) and this action occurs very rapidly, over e period of few minutes. In a range of PaCO2 20mmHg to 80 mmHg the cerebral blood flow changes in a linear manner. End tidal carbon dioxide concentration(EtCO2) is a surrogate measure of PaCO2 (especially in a haemodyanimically stable patient with healthy lungs ) and is routinely monitored continuously in patients subjected to general anaesthesia. To date there is very little literature on the effects changing EtCO2 on ONSD . This prompted us to conduct this study to find out the effects of different levels of EtCO2 on ONSD.

DETAILED DESCRIPTION:
In this study we monitored the effect of three different EtCO2 levels ( 40mmHg,30mmHg and 50mmHg ). In these healthy patients we observed rapid response in ONSD with changes in EtCO2. This again highlights the fact that optic nerve being in direct communication with the brain ,the pressure changes in the latter are reflected in the ONSD. The alteration in ONSD was immediate in response to EtCO2 changes, and moreover,changes in ONSD were parallel to the EtCO2 changes. Since CBF and cerebral blood volume change in response to changes in PaCO2, the ONSD also changes accordingly. Over the years ,advancements in monitoring of ICP has enabled the diagnosis of elevated ICP reliably by non-invasive techniques.Optic nerve sheath diameter measurement using bedside ultrasound has been shown to correlate with clinical and radiologic signs and symptoms of raised ICP. Despite the association between ONSD and PaCO2 , there is scanty literature on ONSD responsiveness to a more dynamic surrogate of PaCO2, that is EtCO2. The pertinent advantages of EtCO2 over PaCO2 measurement is that the former is continuously monitored under anesthesia and avoids time consuming process of arterial blood gas sampling. Moreover, the sensitivity of ICP to even small fluctuations in EtCO2 has been reported in literature. Animal studies have estimated that the rate of this increase in ONSD by 0.0034mm/mmHg increase in ICP.

The ONSD was smallest (0.29cm) at EtCO2 30mmHg, and biggest (0.40cm ) at EtCO2 50mmHg while it was intermediate ( 0.34cm) at EtCO2 40 mmHg. These changes in ONSD are direct representation of changes in ICP brought about by changes in CBF due to PaCO2 changes. Based on results of Bland Altman plots, the calculated 95% confidence interval (CI) for the difference of two measures( EtCO2 40mmHg and 30mmHg ) on ONSD was 0. 009 to 0.102 and the calculated CI for the difference of other two measures ( EtCO2 40mmHg and 50mmHg ) on ONSD was 0.152 to 0. 29 and thus were observed to be statistically insignificant.

Recently Kim et al studied ONSD responsiveness to two levels of EtCO2 ,40 and 50mmHg, each measured at 1 and 5min and they observed significant changes in the diameter of ONSD. Thus their results are at variance with our study. Various possibly reasons for differences in findings are Kim et al studied a small number of patients as opposed to a relatively larger sample size in our study. Also they used total intravenous anesthesia combining propofol and remifentanil infusion. This combination is more likely to predispose patients to systemic hypotension which in turn would increase ICP by causing cerebral vasodilation. Other possibility for different results may be that sonographic measurements of ONSD may vary by the observer's skills or even type of ultrasound device.

According to available literature, the upper limit of ONSD used to define ICP more than 20mmHg (raised ICP ) ranges from 0.48 to 0.57 cm. In our study ,the upper limit of ONSD at EtCO2 level 50mmHg was average of 0.40cm which implies that even at EtCO2 50mmHg, intracranial hypertension is a remote possibility in healthy non-neurosurgical patients with normal brain compliance. We kept constant the factors such as position of patients, time of measurement after achieving target EtCO2, measuring ONSD in a single plain ( transverse) and involving same experienced operator,,thereby, avoiding any confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I adult patients in non head injury category between 18 to 65 years, of either gender undergoing brachial plexus injury surgery under general anesthesia.

Exclusion Criteria:

* Patients with a history of head injury, any respiratory or cardiovascular system disease or non consenting patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All ASA grade I adult patients in non head injury category between 18 to 65 years, of either gender undergoing brachial plexus injury surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Optic nerve sheath diameter [ONSD] measured by ultrasonography in response to change in End tidal Co2 concentration in patients with brachial plexus injury | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Indu Kapoor, Principal Investigator — AIIMS, New Delhi
Locations (1):
- Indu Kapoor, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided